CLINICAL TRIAL: NCT03503604
Title: A Phase Ib Study of hPV19, a Novel Humanized Monoclonal Antibody Against Vascular Endothelial Growth Factor (VEGF),in Combination With Chemotherapy in Patients With Advanced Solid Tumors Refractory to Standard Therapy.
Brief Title: A Study of Anti-VEGF Monoclonal Antibody hPV19 in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SuZhou Stainwei Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STW201701B
Record Dates: First submitted 2018-03-20; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Solid Tumors
Keywords: mAb; VEGF; antibody; phase1
MeSH Terms: interventions — Fluorouracil; Oxaliplatin; Leucovorin; Paclitaxel; Carboplatin; Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Experimental): hPV19 mAb plus FOLFOX(5-Fluorouracil,Oxaliplatin,Leucovorin)
  Interventions: Biological: hPV19 mAb; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin
- group 2 (Experimental): hPV19 mAb plus paclitaxel/carboplatin
  Interventions: Biological: hPV19 mAb; Drug: Paclitaxel; Drug: Carboplatin
- group 3 (Experimental): hPV19 mAb plus gemcitabine/carboplatin
  Interventions: Biological: hPV19 mAb; Drug: Gemcitabine; Drug: Carboplatin
- group 4 (Experimental): hPV19 mAb plus FOLFIRI(5-Fluorouracil,Irinotecan, Leucovorin)
  Interventions: Biological: hPV19 mAb; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Irinotecan

INTERVENTIONS:
Biological: hPV19 mAb — Intravenous (IV) infusions, 4 and 6 milligrams per kilogram (mg/kg) every 2 weeks
  Other Names: anti-VEGF mAb
  Arms: group 1; group 4
Biological: hPV19 mAb — Intravenous (IV) infusions, 6 milligrams per kilogram (mg/kg) every 3 weeks
  Other Names: anti-VEGF mAb
  Arms: group 2; group 3
Drug: 5-Fluorouracil — 400 mg/m2 bolus followed by a 2400 mg/m2 continuous infusion, every 2 weeks
  Arms: group 1; group 4
Drug: Oxaliplatin — IV Infusion, 85 milligrams per square meter (mg/m2) every 2 weeks
  Arms: group 1
Drug: Leucovorin — IV infusion, 400 mg/m2 every 2 weeks
  Arms: group 1; group 4
Drug: Paclitaxel — IV infusion, 175 mg/m2 every 3 weeks
  Arms: group 2
Drug: Carboplatin — IV infusion, AUC=6 every 3 weeks
  Arms: group 2
Drug: Gemcitabine — IV infusion, 1000 mg/m2 at day1 and day 8 every 3 weeks
  Arms: group 3
Drug: Carboplatin — IV infusion, AUC=4 every 3 weeks
  Arms: group 3
Drug: Irinotecan — IV Infusion,180 milligrams per square meter (mg/m2) every 2 weeks
  Arms: group 4

SUMMARY:
hPV19 is a monoclonal antibody (mAb) directed against vascular endothelial growth factor (VEGF). hPV19 binds to human VEGF with unique binding site on VEGF different from that of Bevacizumab(Avastin) and inhibits the binding of VEGF to it's receptors, VEGF-R1 and VEGF-R2. By preventing VEGF binding to its receptors, growth of tumor blood vessels are inhibited and tumor growth prevented or slowed. In this study we are investigating the tolerability, safety, pharmacokinetics and anti-tumor activity of hPV19 in combination with chemotherapy in patients with solid tumors. hPV19 will give to patients by intravenous(i.v.) infusion with a single and multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed malignity
* Measurable disease
* Performance status 2 or less(ECOG)
* Life expectancy ≥3 months

Exclusion Criteria:

* hepatitis C virus (HCV), or HIV antibody positive
* Previously received anti-VEGF mAb or fusion-protein drugs within 28 days nearly
* Evidence of serious infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants That Experienced Any Dose-Limiting Toxicities (DLT) During the DLT Assessment Period | during the first 21 days
  DLTs were adverse events (AEs) possibly related to study drug that met the National Cancer Institute's Common Terminology Criteria for AEs (NCI CTCAE, version 4.03) with any one of the following:
  1. Grade 4 neutropenia ≥7 days; febrile neutropenia; grade 4 anemia; grade 4 thrombocytopenia or grade 3 thrombocytopenia with bleeding;
  2. ≥ grade 3 nonhematologic toxicity with the exception of nausea, vomiting, diarrhea, dehydration or electrolyte abnormalities that resolved to a lower grade with maximum supportive treatment within 3 days;
  3. ≥Grade 3 hypertension that cannot resolved to a lower grade with supportive treatment within 2 weeks or uncontrolled hypertension;
  4. Urine protein ≥3.5 grams/24 hours and cannot resolved to < 1.0 grams/24 hours within 2 weeks;
  5. Gastrointestinal perforation: symptoms, signs and imaging evidence of abdominal pain require surgical treatment;
  6. Grade 3 or 4 arterial thromboembolism, including stroke and myocardial infarction;
Number of Participants With hPV19 Drug-Related Adverse Events or Serious Adverse Events | Baseline to the last dose plus 28 days.
  Data are presented for the number of participants who experienced treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), Grade ≥3 TEAEs, or adverse events (AEs) leading to discontinuation of treatment that were considered to be related to hPV19. Events related to chemotherapy were reported separately.

SECONDARY OUTCOMES:
Number of Participants With Serum Anti-hPV19 Antibodies (Immunogenicity) | before Single dose; Day 21 of 21-day DLT assessment period; Every 8 or 9 weeks after 21-day DLT assessment period.
Maximum Concentration (Cmax) of hPV19 | Single dose(Cycle 1)：2h before administered; after administered 10min±5min、4h±30min、24h±1h、168h±1h、336h±1h. Other cycles: 2h before administered and after administration 10min±5min.
Area Under the Curve (AUC) of hPV19 | Single dose(Cycle 1)：2h before administered, after administered 10min±5min、4h±30min、24h±1h、168h±1h、336h±1h. Other cycles: 2h before administered and after administration 10min±5min.
Half Life (t1/2) of hPV19 | Single dose(Cycle 1)：2h before administered, after administered 10min±5min、4h±30min、24h±1h、168h±1h、336h±1h. Other cycles: 2h before administered and after administration 10min±5min.
  t1/2 is the time required for the plasma/serum concentration to decrease 50%
Clearance (CL) of hPV19 | Single dose(Cycle 1)：2h before administered, after administered 10min±5min、4h±30min、24h±1h、168h±1h、336h±1h. Other cycles: 2h before administered and after administration 10min±5min.
Steady State Volume of Distribution (Vss) of hPV19 | Single dose(Cycle 1)：2h before administered; after administered 10min±5min、4h±30min、24h±1h、168h±1h、336h±1h. Other cycles: 2h before administered and after administration 10min±5min.
  Vss is the theoretical volume in which the total amount of study drug would need to be uniformly distributed during steady state to produce the same concentration as it is in plasma/serum
Best Overall Response [Anti-Tumor Activity of hPV19 Plus Chemotherapy] | Up to six months after 1st treatment or until progression of disease (PD)
  Best overall response evaluated using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria.
  Complete Response (CR): disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). Partial Response (PR): at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. Progressive Disease (PD): an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if that was the smallest on study). In addition, the sum must have demonstrated an absolute increase of at least 5 mm (the appearance of 1 or more new lesions was considered progression). Stable Disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China